CLINICAL TRIAL: NCT05251818
Title: Effect of Acupressure on Bowel Functions After Cesarean Section: A Randomized Controlled Trial
Brief Title: Effect of Acupressure on Bowel Functions After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, resmiye kaya odabaş, Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Resmiye-03
Record Dates: First submitted 2022-02-03; First posted 2022-02-23 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Acupressure; Bowel Functions
Keywords: Acupressure; Bowel movemet; Caaesarean sectio; Defecation; Flatulence.
MeSH Terms: conditions — Flatulence | interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure grubu (Active Comparator): The first thing after the operation is to apply the thumb tool for approximately seven minutes, with 15 seconds of preparation and 1.5 minutes of application at each point of the LI4 and TH6 acupuncture points (the equivalent of working each point).The second application will be repeated three hours after the first application, with the same procedure.
  By the researcher, hourly monitoring will be done until the bowel sounds of the puerperant are heard, and the puerperant will be followed up until the gas and defecation output. The gas and defecation time of the puerperants will be questioned every 12 hours, and the information will be obtained by making a phone call with those who are discharged without defecation.
  Interventions: Other: acupressure
- Control Group (Active Comparator): No application will be made to the control group.. From the first postoperative hour, the researcher will follow the bowel sounds every hour until the first bowel sounds of the patient are heard.
  Postpartum women will be followed until gas and defecation are released. The gas and defecation time of the puerperants will be questioned every 12 hours, and the information will be obtained by making a phone call with those who are discharged without defecation.
  Interventions: Other: Control

INTERVENTIONS:
Other: acupressure — A suitable environment will be prepared for postpartum women where privacy can be protected. Application points will be determined by choosing the most comfortable position of the mother. LI4 and TH were selected as the most preferred points among the points reported to be effective on intestinal functions by scanning the literature on the determined points. Acupressure will be applied to the LI4 and TH6 points for a total of 12 minutes in the first hour after the surgery. Light pressure will be applied with the thumb of the practitioner's hand. After applying pressure for 2 minutes for each point, it is passed to the other point in the symmetrical region and the application is done without interruption
  Arms: Acupressure grubu
Other: Control — No application will be made to puerperant women in this group. Only hourly follow-up will be done until the first bowel sound is heard. In addition, defecation and gas extraction will be questioned every 12 hours.
  Arms: Control Group

SUMMARY:
Enema application to pregnant women and prohibition of oral feeding before cesarean section, general anesthesia applied during cesarean section, pain in the post-cesarean period, limitation of movement, insufficient fluid intake, low-fiber diet, hospital environment and drugs such as narcotics cause constipation. In addition, one of the most common complications after abdominal surgeries is postoperative ileus. Many noninvasive applications help to overcome this problem. This study was planned as a randomized controlled trial to examine the effect of acupressure on bowel functions after cesarean section. The research will be carried out between July 2021 and July 2022 at the Samsun Training and Research Hospital Gynecology and Pediatrics Hospital affiliated to the Samsun Provincial Health Directorate. The research will be carried out with two groups as acupressure and control group. The sample number was calculated using the G*Power 3.1.9.2 program and the acupressure group: 26 and the control group: 26. In order to increase the analysis power, the number of people for each group was taken as 30 (n=60). It is planned to collect the data with the Postpartum Information Form. After the women in the acupressure group come to the service, 2 applications will be made in the first postpartum hour and 3 hours after the first application, and no application will be made to the control group. Intestinal sounds will be monitored every hour until the first bowel sounds are heard, and the "Postpartum Registration Form" given to the woman will be received and recorded at the post-op 24th hour. The data of the research will be evaluated using the Statistical Package for the Social Sciences 22.0 program. In the evaluation of the data; descriptive statistics percentage, arithmetic mean±standard deviation, median and minimum-maximum values will be given. Student t test, ANOVA test will be used for those with normal distribution, Mann-Whitney U and Kruskal Wallis tests for those who are not. Type 1 error level will be taken as 0.05. Pearson Correlation test will be applied to determine the relationship between the intestinal functions of the experimental group and the tests. Statistical significance level will be accepted as p<0.05

DETAILED DESCRIPTION:
H01: There is no difference between the acupressure and control groups in terms of hearing time of bowel sounds.

H02: There is no difference in gas removal time between acupressure and control groups.

H03: There is no difference between the acupressure and control groups in terms of time to defecation.

This study was designed as a randomized controlled experimental study. The study will be carried out between July 2021 and July 2022 in the "Samsun Training and Research Hospital Gynecology and Pediatrics Hospital gynecology service".The universe of the research will be women who gave cesarean section under general anesthesia in Samsun Training and Research Hospital, Gynecology and Pediatrics Hospital.

The G-Power program was used to determine the sample of the study and it was planned to recruit 60 women in total (acupressure group: 30 women, control group: 30 women). The data of the research will be collected with the Postpartum Information Form created by the researcher. Which group the participants will be in will be determined by the full randomization technique on the website www.randomizer.org. After obtaining the permission of the ethics committee and the institution to carry out the study, the women who had a cesarean section will be met by going to the institution. Mothers who meet the research criteria will be informed about the purpose, content and methods of the research, and verbal and written consent will be obtained from those who want to participate. The researcher will fill in the "Postpartum Information Form" by interviewing the pregnant women face-to-face before the cesarean section, examining their socio-demographic and obstetric characteristics, and the operation information from the patient's file after the cesarean section.

Postpartum Information Form: This form was developed by researchers based on the literature. It consists of questions that include socio-domographic and obstetric characteristics and surgical information. Within the scope of the research, 7 questions including socio-demographic characteristics of pregnant women (age, education level, occupation, amount of fluid intake, economic status, bowel habits before and during pregnancy), 8 questions including obstetrical characteristics (gestational week, number of pregnancies, number of abortions, miscarriage) number of children, number of living children, number of live births, previous type of delivery, reason for cesarean section), 7 questions including surgery information (time of start and end of surgery, fasting time before surgery, total amount of fluid given during surgery, amount of blood lost during surgery, admission to the ward). date and time, bowel function status of women after surgery) consists of a total of 22 questions.

Pre-Application In order to assess whether the questions have been understood, a preliminary study will be conducted with five mothers before starting the study. As a result of the evaluation, it will be evaluated whether there is a need for editing in the data forms and adjustments will be made. Those included in the preliminary study will not be included in the sample group.

Data Collection After acupressure, the woman will be ready to serve. The control process will be any application.

A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position for the mother, leaving the application points open. The most preferred points on intestinal functions were LI4 and TH6 points. LI4 (Hegu) and TH6 pressure points will be applied consecutively. Depending on the preparation and compression time on the 2 selected points (4 points with each point on the other extremity), the session duration of an individual will be approximately 12 minutes. While practicing, the researcher will check the time using a digital wristwatch with a stopwatch.

LI4: It is the point where the cambered muscle group is when the thumb and forefinger are brought closer together. In other words, it corresponds to the midpoint of the metacarpal bone of the index finger. This area is often preferred for problems such as face, head, toothache, stomachache, abdominal pain, constipation, diarrhea, dysentery, dysmenorrhea, amenorrhea, difficult or abnormal birth.

TH 6: Located on the outer side of the arm, 4 fingers above the wrist crease, on the midline of the arm (between radius and ulna bones).

This point is used in the treatment of constipation, irritable colon disease, hoarseness.

First, after 2 minutes of pressure is applied to the LI4 compression point on both hands, the TH 6 compression point on both arms will be applied consecutively without interruption. Although there is a difference in the order of use of the determined acupressure points, in this study, first LI4 and then TH 6 points will be performed. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch. The practitioner has acupressure training on this subject.

Analysis of Data The data of the study will be evaluated using the Statistical Package for the Social Sciences (SPSS) 22.0 program. All data will first be evaluated with Kolmogorov-Smirnov for conformity to normal distribution and then analyzed according to fitness for normal distribution. For descriptive statistics, percentages will be used in general, arithmetic mean±standard deviation for those suitable for normal distribution, median and minimum-maximum values for those that do not fit. In the analysis of the data, student t test and ANOVA test will be used for those with normal distribution, and Mann-Whitney U and Kruskal Wallis tests for those who do not. Type 1 error level will be taken as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* Having a cesarean section with general anesthesia,
* After the operation, non-narcotic and the same type of analgesic substance is applied to provide pain control,
* Able to speak and understand Turkish,
* Postpartum women with at least primary school graduates will be included in the study.

Exclusion Criteria:

* Being obese (BMI≥30),
* Opioid medication given in the post-op period,
* Any disease related to the digestive system,
* Having a history of abdominal surgery,
* Chronic constipation or irregularity in defecation habits,
* Having any chronic disease (such as diabetes, hypertension, heart failure),
* Pregnancy complications (such as preeclampsia, gestational diabetes),
* The baby is in the intensive care unit,
* Having any physical problem that will prevent the application of acupressure to LI4 and TH 6 points,
* Women who develop disorders or insufficiency related to fluid-electrolyte balance, acid-base balance and tissue perfusion during and after the operation will not be included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
First bowel sound | until the first bowel sound to 24 hours
  Bowel sounds will be heard from the abdominal region of the woman with a stethoscope every hour.
Gas removal time | until the first gassing up to 24 hours
  Hourly follow-up until the first gas removal time is heard
Time to defecate | First defecation up to one week after cesarean section
  Questioning every 12 hours until the first stool output

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Sökmen, Lectur, Principal Investigator — Ondokuz Mayıs University; Resmiye Kaya Odabaş, Ress. Ass., Study Chair — Kocaeli University University; Ayten Taşpınar, Prof. Dr., Study Chair — Aydin Adnan Menderes University
Locations (1):
- Samsun Training and Research Hospital Gynecology and Pediatrics Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No